CLINICAL TRIAL: NCT02727231
Title: Closing the Loop in Adults With Type 1 Diabetes and HbA1C<7.5% Under Free Living Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Dr Roman Hovorka, Dr, University of Cambridge
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AP@home04 phase2
Record Dates: First submitted 2016-03-29; First posted 2016-04-04 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Type 1 Diabetes
Keywords: closed loop glucose control; hypoglycemia; type 1 diabetes; HbA1C<7.5%
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- day and night closed loop control (Experimental): Subjects glucose levels are controlled by Florence D2A or similar closed loop insulin delivery system
  Interventions: Device: Florence D2A or similar closed loop glucose control system
- usual insulin pump therapy management (Active Comparator): Subject glucose level controlled by usual insulin pump therapy in conjunction with continuous glucose monitoring (FreeStyle Navigator CGM)
  Interventions: Device: CSII with CGM

INTERVENTIONS:
Device: Florence D2A or similar closed loop glucose control system — Subject's glucose level will be controlled by the Florence D2A or similar automated closed loop glucose control system. The system comprises of FreeStyle Navigator 2 ® Continuous Glucose Monitoring (CGM) System (Abbott Diabetes Care, Alameda, CA, USA), Dana R Diabecare subcutaneous insulin infusion pump (Sooil Corp. Seoul, South Korea)or similar insulin pump, and MPC-based glucose control algorithm running on a smartphone
  Arms: day and night closed loop control
Device: CSII with CGM — Subject glucose level controlled by usual insulin pump therapy in conjunction with continuous glucose monitoring (CGM)
  Arms: usual insulin pump therapy management

SUMMARY:
The main objective of this study is to determine whether day and night closed-loop insulin delivery for 4 weeks under free living conditions is superior to usual insulin pump therapy in adults with type 1 diabetes and HbA1C<7.5%.

This is an open-label, multi center, randomized, crossover design study, involving a 2-4 week run-in period, followed by two 4 weeks study periods during which glucose levels will be controlled either by an automated day- and night closed-loop system or by subjects usual insulin pump therapy in random order. A total of up to 34 adults (aiming for 24 completed subjects) aged 18 years and older with T1D on insulin pump therapy and HbA1C<7.5% will be recruited through diabetes clinics and other established methods in participating centers.

Subjects will receive appropriate training in the safe use of closed-loop insulin delivery system. Subjects will have regular contact with the study team during the home study phase including 24/7 telephone support.

The primary outcome is time spent in target range between 3.9 and 10.0 mmol/L as recorded by CGM during home stay. Secondary outcomes are time spent with glucose levels above and below target, as recorded by CGM, and other CGM-based metrics.

ELIGIBILITY:
Inclusion Criteria:

* The subject has type 1 diabetes as defined by WHO
* The subject is 18 years of age or older
* The subject will have been on an insulin pump for at least 6 months with good knowledge of insulin self-adjustment including carbohydrate counting
* The subject is treated with one of the rapid acting insulin analogues (Insulin Aspart, Insulin Lispro or Insulin Glulisine)
* HbA1c <7.5% (58mmol/mmol) based on analysis from central laboratory or equivalent
* The subject is willing to perform regular finger-prick blood glucose monitoring, with at least 6 measurements per day
* The subject is willing to wear closed-loop system at home and at work place
* The subject is willing to follow study specific instructions
* The subject is willing to upload pump and CGM data at regular intervals
* Female subjects of child bearing age should be on effective contraception and must have a negative urine-HCG pregnancy test at screening.

Exclusion Criteria:

* Non-type 1 diabetes mellitus
* Any other physical or psychological disease or condition likely to interfere with the normal conduct of the study and interpretation of the study results
* Current treatment with drugs known to have significant interference with glucose metabolism, such as systemic corticosteroids, as judged by the investigator
* Known or suspected allergy against insulin
* Subjects with clinically significant nephropathy, neuropathy or proliferative retinopathy as judged by the investigator
* Significantly reduced hypoglycaemia awareness as judged by the investigator
* More than one episode of severe hypoglycaemia as defined by American Diabetes Association in preceding 6 months (Severe hypoglycaemia is defined as an event requiring assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions).
* Random C-peptide > 100pmol/l with concomitant plasma glucose >4 mM(72 mg/dl) Total daily insulin dose > 2 IU/kg/day
* Subject is pregnant or breast feeding or planning pregnancy in near future (within next 3 months)
* Severe visual impairment
* Severe hearing impairment
* Subjects using implanted internal pacemaker
* Lack of reliable telephone facility for contact
* Subject not proficient in English (UK) or German (Austria)
* Subjects who are living alone
* Additional exclusion criteria specific for Austria: Positive results on urine drug screen (amphetamines/metamphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates).
* Additional exclusion criteria specific for Austria:Positive alcohol breath test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-03; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Time spent in the target glucose range (3.9 to 10.0 mmol/l) based on subcutaneous glucose monitoring | 4 weeks
  Time spent in the target glucose range from 3.9 to 10.0 mmol/l based on subcutaneous glucose monitoring (CGM) during the 4 weeks of home stay. Intention to treat basis.

SECONDARY OUTCOMES:
Continuous subcutaneous glucose monitoring (CGM) based outcome | 4 weeks
  Time spent above and below the target glucose range from 3.9 to 10.0 mmol/l based on subcutaneous glucose monitoring (CGM) during the 4 weeks of home stay. Intention to treat basis.
Continuous subcutaneous glucose monitoring (CGM) based outcome | 4 weeks
  Average,standard deviation and coefficient of variation of glucose levels during 4 weeks of home periods
Continuous subcutaneous glucose monitoring (CGM) based outcome | 4 weeks
  The time with glucose levels < 3.5 mmol/l and <2.8 mmol/l during 4 weeks of home periods
Continuous subcutaneous glucose monitoring (CGM) based outcome | 4 weeks
  The time with glucose levels in the significant hyperglycaemia,(glucose levels > 16.7 mmol/l during 4 weeks of home periods
Continuous subcutaneous glucose monitoring (CGM) based outcome | 4 weeks
  Low Blood Glucose Index
Continuous subcutaneous glucose monitoring (CGM) based outcome | 4 weeks
  The "Area Under the Curve" below 3.5 mmol/l during 4 weeks home periods
Continuous subcutaneous glucose monitoring (CGM) based outcome | 4 weeks
  Between 24 hour period variability: Coefficient of variation of CGM glucose between 24 hour periods (midnight to midnight)
Continuous subcutaneous glucose monitoring (CGM) based outcome during overnight period between 24:00 and 06:00 | 4 weeks
  Time spent with CGM glucose concentration in range 3.9-10.0mmol/L
Continuous subcutaneous glucose monitoring (CGM) based outcome during day period between 06:00 to 24:00 | 4 weeks
  Time spent with CGM glucose concentration in the target range (3.9-10.0mmol/L)
Insulin dose | 4 weeks
  Total, basal and bolus insulin dose during 4 weeks of home periods
Adverse Events | 5 months
  Safety evaluation will comprise the number of episodes of hypoglycaemia, significant ketonemia (> 3.0mmol/l)as well as nature and severity of any other adverse events
Utility Evaluation | 4 weeks
  Utility evaluation is the percentage of closed-loop operation time during use at home, and when CGM was available

OTHER OUTCOMES:
Accuracy of CGM | 4 weeks
  CGM accuracy during 4 weeks home period; Capillary glucose vs. CGM will be evaluated using standard measures of numerical and clinical accuracy including absolute relative deviation and error grid analysis

CONTACTS AND LOCATIONS:
Overall Officials: Roman Hovorka, Principal Investigator — University of Cambridge
Locations (2):
- Medical University of Graz, Graz, Austria
- Cambridge University Hospitals NHS Foundation Trust, Addenbrookes Hospital, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- [Derived] Bally L, Thabit H, Kojzar H, Mader JK, Qerimi-Hyseni J, Hartnell S, Tauschmann M, Allen JM, Wilinska ME, Pieber TR, Evans ML, Hovorka R. Day-and-night glycaemic control with closed-loop insulin delivery versus conventional insulin pump therapy in free-living adults with well controlled type 1 diabetes: an open-label, randomised, crossover study. Lancet Diabetes Endocrinol. 2017 Apr;5(4):261-270. doi: 10.1016/S2213-8587(17)30001-3. Epub 2017 Jan 14. PMID 28094136